CLINICAL TRIAL: NCT03267953
Title: Adaptive Internet-based Stress Management Among Adults With a Cardiovascular Disease: A Pilot Sequential Multiple Assignment Randomized Trial (SMART) Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Mary's Research Center, Canada (Other)
Collaborators: McGill University (Other)
Responsible Party: Principal Investigator, Sylvie Lambert, Assistant professor, McGill University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: SMHC 17 11
Record Dates: First submitted 2017-08-28; First posted 2017-08-31 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: Cardiovascular Diseases; Stress, Psychological
Keywords: Stress management, e-Health, cardiovascular disease, adaptive design, lay coaching, motivational interviewing
MeSH Terms: conditions — Cardiovascular Diseases; Stress, Psychological | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First stage: Self-directed My Health CheckUp (Experimental): Participants randomized to this group will be sent an e-mail invitation by the research team to register to the website. Once registered, participants will receive a second e-mail that will provide brief instructions on getting started and invite them to use the website for 12 weeks ad libitum. No additional contact will be provided thereafter by research team.
  Interventions: Behavioral: My Health CheckUp Online Stress Management Program
- First stage: Minimally guided My Health CheckUp. (Experimental): This group will also be invited to use the 12-week Internet-based stress management program, but they will additionally receive support via weekly telephone calls from a lay coach.
  Interventions: Behavioral: My Health CheckUp Online Stress Management Program; Behavioral: Lay telephone coaching
- Second stage: High intensity Motivational Interviewing (MI) (Experimental): After 6 weeks, response to the first stage programs will be assessed and only the non-responders will be randomized a second time to (a) continue with the first stage programs or (b) High-intensity MI. In addition to continued access to My Health CheckUp, participants in this group will also be supported with 6 weekly, telephone-based MI sessions.
  Interventions: Behavioral: My Health CheckUp Online Stress Management Program; Behavioral: Motivational interviewing (telephone)

INTERVENTIONS:
Behavioral: My Health CheckUp Online Stress Management Program — Self-contained, web-based, stress management program developed by team of health care professionals, designed to encourage patients to learn evidence-based cognitive and behavioural strategies to effectively manage stress. Health risk appraisals include evidence-based recommendations to address risks. Stress management modules include education about the impact of stress, self-monitoring through a stress diary, and using four key strategies: physical activity, deep breathing and relaxation, problem-solving/addressing negative thoughts, and sleep hygiene. Through the modules, patients will learn new stress management strategies and have an opportunity to practice these, track their progress, and obtain feedback via the website. To facilitate self-monitoring of stress levels and tracking of strategies such as physical activity, tracking tools can be used on mobile devices.
Behavioral: Lay telephone coaching — The goal of telephone coaching will be to provide brief encouragement on how to use the modules; however, no formal therapy will be provided. Sessions will range between 10-15 minutes. Each coach session will follow the process outlined by the GROW model, which stands for Goal, Reality, Options/Obstacles, and Will/Way forward. The sessions will start with the coach and participant agreeing on the topics for discussion and desired outcomes (goal). Then, coaches will explore the use of the intervention over the previous week, guide participants through the modules, identify barriers to using these modules, offer advice to overcome these barriers, and provide positive reinforcement. The development of an action plan for the following week will conclude each session. The short Perceived Stress Scale will be used at the end of each session to monitor progress. A script will guide the lay coach through each call.
  Arms: First stage: Minimally guided My Health CheckUp.
Behavioral: Motivational interviewing (telephone) — Sessions will range from 30 to 45 minutes. The goal of MI is to strengthen patients' motivation and confidence for adopting the stress management strategies suggested. The MI practitioner's interventions are based on the four processes of MI: Engaging, Focusing, Evoking, and Planning.
  Arms: Second stage: High intensity Motivational Interviewing (MI)

SUMMARY:
Internet-based stress management programs adapted to patients' needs

Stress is inevitable, and it has many negative consequences on the health of everybody, but particularly on the health of patients with a cardiovascular disease (CVD). The good news is that patients with CVD can learn to better control their stress through stress management programs. Most stress management programs are offered face-to-face by a trained health care professional. Research has shown that these programs have a positive impact on the health of patients with CVD, including reducing mortality and other risk factors that can make the disease worse (e.g., reduces blood pressure). Because of these benefits, the recommendation is to offer a stress management program to as many patients with CVD as possible. The problem is that their delivery is challenging for most clinics (e.g., too costly to run, health care professionals are not available). This means many good stress management programs never make it to the patient. Patients also face barriers in accessing traditional stress management programs such as stigma or need to travel. Therefore, new approaches are needed to allow findings from research to actually have an impact on the public's health.

One of these approaches is to use the internet to deliver stress management programs. The internet has now been used for about 10 years to deliver a range of programs to patients. There are limitations to this approach as well. For instance, 40-60% of patients who will use an internet-based program will not benefit from it. These patients need more support or guidance to get the most out of their internet-based program. This is the problem addressed using the proposed innovative trial design. Investigators aim to improve the number of patients with CVD who improve after receiving a stress management program by changing the type and level of support they receive over time. This type of innovative trial design is more and more popular, but has never been used to enhance a stress management programs for patients with CVD.

DETAILED DESCRIPTION:
BACKGROUND: Stress has a negative impact on the experience of individuals with a cardiovascular disease-both directly (e.g., physiologic effects of stress may worsen cardiovascular disease) and indirectly (e.g., leads to higher perceived symptom severity). Therefore, stress management has become an extensively researched form of psychological therapy for these individuals, and is increasingly offered through the internet. Advantages of internet-based interventions include being time efficient (e.g., cut travel time), reducing waiting-lists, and increasing access for some sub-groups of the population (e.g., those living in rural and remote areas). Internet-based interventions also have the potential to integrate effective features of face-to-face interventions (e.g., tailored feedback, monitoring), but offer the scalability needed for public health interventions. However, up to 60% of individuals do not respond to these interventions, and for these individuals offering different types of support or increasing the intensity of the support provided is necessary. An innovative trial design to develop time-varying, adaptive interventions to maximize clinical effectiveness is the Sequential multiple assignment randomized trials (SMARTs). However, despite increasing popularity, SMARTs remain relatively new to intervention researchers.

GOAL AND OBJECTIVES: The goal of this pilot Sequential Multiple Assignment Randomized Trial (SMART) is to inform the planning of a subsequent larger SMART to evaluate an adaptive internet-based stress management program that follows a stepped-care model for adults with a cardiovascular disease. The primary objectives are to examine the (a) feasibility of the SMART procedures and different combinations of the stress management program (recruitment, retention, and questionnaire completion rates, reach, and fidelity) and (b) acceptability of the combinations of the stress management program, including adapting the program for non-responders and assessing adherence, satisfaction, and stress management strategies learned. The secondary objective is to estimate the program's effect size to inform sample size calculations for a full-scale SMART.

METHODOLOGY: 56 patients with a physician confirmed diagnosis of a cardiovascular disease will be recruited through clinic referrals and community-based study advertisement. Inclusion criteria are: (a) moderate stress (stress subscale score of 15 or more on Depression, Anxiety, and Stress Scale), (b) at least 18 years of age, (c) not participated in a stress management intervention in the past year, (e) regular access to a computer with internet and e-mail capabilities, and (f) reports understanding English or French. Eligibility will be confirmed mainly by self-report at the time of a screening interview. After completing their consent form and baseline questionnaire (T0), participants will be randomized to either: (a) a 6-week self-directed, web-based stress management program or (b) the same program plus weekly lay coaching. At the end of 6 weeks, intervention response will be assessed (T1 questionnaire), and non-responders will include those who have a stress score that did not improve (i.e., less than 50% decrease) or have a stress score above the cut-off point for mild stress (primary tailoring variable). In both groups, non-responders will then be randomized a second time to either (a) continue with their first stage program or (b) professionally-led motivational interviewing for another 6 weeks. During this time, responders will continue their first stage programs. The internet-based stress management program is available through my Health CheckUp. All participants will then complete their 12-13 weeks follow-up questionnaire (T2) to examine changes in stress and quality of life (primary outcomes), anxiety, depression, illness appraisal, self-efficacy, physical activity, and coping (secondary outcomes). Acceptability will be assessed by the satisfaction measure included in the follow-up questionnaire and further explored during an exit interview with participants. Feasibility measures will focus on the characteristics of the participants reached, protocol fidelity, percent of missing data, and recruitment and retention rates.

SIGNIFICANCE: The potential reach of internet-based interventions promises considerable public health impact. However, to maximize impact, the most effective interventions need to be developed and adapted to patients' evolving needs. This study will use the innovative SMART design to evaluate an adaptive internet-based intervention for individuals with a physical chronic illness.

ELIGIBILITY:
Inclusion Criteria:

* physician-confirmed diagnosis of a CVD (at least 3 months since most recent diagnosis)
* moderate stress as indicated by a score of > 15 on the stress subscale of the Depression, Anxiety, and Stress Scale (DASS)
* regular access to a computer with Internet and e-mail capabilities
* understands English or French

Exclusion Criteria:

* participated in a stress management program in the past year
* hospitalized or living in a long-term care residence
* moderate-severe cognitive impairment (Blessed Orientation-Memory-Concentration test score 10+)
* severe stress (DASS stress score > 34)
* suicidal intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Feasibility | Recruitment over 6 months, participant follow-up over 13 weeks
  defined as the practicality of implementing the SMART procedures and of offering different types and levels of support in conjunction with an Internet-based stress management program. Feasibility measures include fidelity, reach, recruitment rate, and questionnaire completion rates.
Acceptability | Recruitment over 6 months, participant follow-up over 13 weeks
  defined as patients' views of the programs, and will include satisfaction with the different types of support offered, appropriateness of adapting the programs for non-responders, examining attrition, and assessing adherence and skills learned.

SECONDARY OUTCOMES:
Clinical significance | At T2: 12-13 weeks
  clinical significance of adapting the type and level of support provided on the primary and secondary outcomes of interest.

OTHER OUTCOMES:
Stress | At T0 (Baseline), T1 (6 weeks) and T2 (12-13 weeks)
  Measured with the Depression, Anxiety, and Stress Scale
Quality of life | At T0 (Baseline), T1 (6 weeks) and T2 (12-13 weeks)
  Measured with the SF-12

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie D Lambert, PhD, Principal Investigator — McGill University
Locations (1):
- St Mary's Hospital Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No